CLINICAL TRIAL: NCT05400239
Title: SOTO Study: Prospective Study to Correlate the Treatment Sensitivity of Patient-derived Organoids With Clinical Outcomes in Head and Neck Squamous Cell Carcinoma (HNSCC) Patients
Brief Title: SOTO: Treatment Sensitivity of Organoids to Predict Treatment Outcome
Status: Recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SOTO Study 305689
Record Dates: First submitted 2022-04-20; First posted 2022-06-01 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Head and Neck Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Surgically resectable disease, followed by adjuvant radiotherapy +/- chemotherapy
- Cohort 2: Primary radiotherapy +/- concurrent chemotherapy
- Cohort 3: Recurrent or metastatic HNSCC undergoing platinum based chemotherapy +/- cetuximab

SUMMARY:
In this study, we aim to assess whether Patient Derived Organoids can be used to predict treatment sensitivity in HNSCC patients.

DETAILED DESCRIPTION:
This is a prospective observation study to generate patient-derived organoids from patients' samples to assess treatment response and to correlate with patients' treatment outcomes and to collect preliminary data on the ability of PDOs to predict patients' treatment response and whether their radiosensitivity and chemosensitivity can be correlated with their survival outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck squamous cell carcinoma (including oral cavity, oropharynx, paranasal sinuses, hypopharynx or larynx) undergoing curative treatment (primary surgery or radiotherapy) or presenting with recurrent or metastatic cancers
* Age > 18 years old

Exclusion Criteria:

* Patients unable to give informed consent e.g. mental disability or vulnerable adults

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a prospective study with a one-year pilot study aiming to recruit 20 patients, which is the realistic target for year 1. The results from year 1 will be used to estimate the sample size for future prospective observation study
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Successful Organoids | 1 Year
  To assess the percentage of successful generated organoids from tissues in head and neck cancer patients

SECONDARY OUTCOMES:
Sensitivity | 1 Year
  To assess the sensitivity of radiotherapy, platinum (cisplatin and/or carboplatin) chemotherapy or cetuximab or their combination in PDOs
Treatment Outcome | 1 Year
  To correlate the treatment sensitivities of PDOs with the treatment outcome of patients

OTHER OUTCOMES:
Treatment Sensitivities | 1 Year
  To correlate the treatment sensitivities of PDOs with the detection rates of plasma ctDNA (all cohorts)
Patients Features | 1 Year
  To assess and correlate the histopathological, genomic and transcriptomic features of patients' samples with PDOs
PDOs Sensitivities | 1 Year
  To assess the sensitivities of PDOs to various targeted therapies based on their genomic profiles
Translational Research | 1 Year
  Collection of archival tissues, blood samples (for ctDNA and PBMC), saliva (for ctDNA), urine or stool samples for other translational research

CONTACTS AND LOCATIONS:
Locations (1):
- Guys Hospital, London, United Kingdom

REFERENCES:
- [Derived] Vasiliadou I, Cattaneo C, Chan PYK, Henley-Smith R, Gregson-Williams H, Collins L, Wojewodka G, Guerrero-Urbano T, Jeannon JP, Connor S, Davis J, Pasto A, Mustapha R, Ng T, Kong A. Correlation of the treatment sensitivity of patient-derived organoids with treatment outcomes in patients with head and neck cancer (SOTO): protocol for a prospective observational study. BMJ Open. 2024 Oct 10;14(10):e084176. doi: 10.1136/bmjopen-2024-084176. PMID 39389599

DOCUMENTS (1):
  • Study Protocol (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT05400239/Prot_000.pdf